CLINICAL TRIAL: NCT00580450
Title: Phase I/II Clinical Trial on Thymosin Alfa 1 of Allogeneic Hematopoietic Transplantation
Brief Title: Thymosin Alfa 1 in Recipients of Allogeneic Hematopoietic Transplantation for Hematological Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Andrea Velardi, Hematology Section, University of Perugia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (ST 1472); ST 1472 06/01/27
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-11

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Thymalfasin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (No Intervention)
- 1 (Experimental)
  Interventions: Drug: Thymosin alpha 1

INTERVENTIONS:
Drug: Thymosin alpha 1 — 1.6 mg sc once a day for 16 weeks
  Arms: 1

SUMMARY:
The purpose of this trial is to determine safety and efficacy of 16 weeks treatment with thymosin alpha 1 given at 1.6 mg dose once daily by subcutaneous injection in adult patients with hematological undergone allogenic bone marrow transplantation and CMV positive.

The efficacy will be explored assessing the ability of thymosin alpha1 to prevent the infection complications.

DETAILED DESCRIPTION:
This is an open label, monocenter, explorative study . A total of 9 patients will be included in the study in three sequential cohort of 3 patients each. Patients will enter into the study after meeting the inclusion and exclusion criteria and signing the Informed Consent Form.

The first three patients will be treated for 16 weeks starting 40 days after transplantation; if all three patients will complete the treatment period without any serious treatment related adverse event then the recruitment of second cohort of patients will be opened and patients treated starting from 20 days after transplantation. The same procedure will be applied for the third cohort of patients starting treatment from day of transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age > 18 or < 55.
3. Patients with AML, ALL, or other haematological malignancies with an indication to transplant with or without a matched donor undergoing allogenic haploidentical hematopoietic transplantation (see Appendix 2) in any of the following categories:

   * Patients in first complete remission (CR) at high risk of relapse because of unfavourable cytogenetics, such as:

     * t (9;22)
     * 11q23 translocation
     * complex karyotype
     * t (8;12)/ETV6-AML
     * t (6;9)/DEK-CAN
     * t (11;14)(q15,q11)
     * Trisomy 13
     * FLT-3/ITD
   * Or other adverse prognostic factors, such as:

     * Secondary leukemia
     * CR after second line treatment
     * High blast count
     * Biphenotypic leukemia
   * Patients in 2nd or 3rd CR or in chemoresistant relapse
4. Recipient CMV positive as measured by pp65 antigenemia and PCR
5. Adequate cardiac function: Asymptomatic of if symptomatic then left ventricular ejection fraction at rest be >45% and must improve with exercise,
6. Adequate hepatic function: <2 x GOT and GPT and <2.0 mg total serum bilirubin unless liver is involved in disease,
7. Adequate renal function: Serum creatinine within normal range or if serum creatinine outside normal range then creatinine clearance >50 ml/min,
8. Adequate Pulmonary function: Diffusion capacity >50% of predicted (corrected for hemoglobin)
9. Normal TSH or evidence of proper thyroid hormone replacement.
10. For women of childbearing potential participating in the study, abstinence from sexual intercourses or use of a reliable form of effective contraception during the treatment period. These may include, but are not limited to, birth control pills, IUDs, condoms, diaphragms, implants, surgical sterilization, or being in a post-menopausal state.
11. Negative pregnancy test prior to first study medication dose.

Exclusion Criteria:

1. Evidence of active hepatitis (B and/or C) or cirrhosis
2. HIV positive
3. Presence of any other active, uncontrolled bacterial, viral or fungal infection
4. Neurological or psychiatric dysfunctions which would impair compliance with the medical regimens and/or transplantation toleration
5. Concomitant or prior history of malignancy other than surgically cured in situ carcinoma of the cervix.
6. Pregnancy as documented by a urine pregnancy test or lactation.
7. Any indication that the patient would not comply with the conditions of the study protocol.
8. Previous treatment with thymosin alpha 1.
9. Simultaneous participation in another investigational drug study or participation in any clinical trial involving investigational drugs within 3 months before study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2007-12; Primary Completion 2007-12 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of improvement of immunological reconstitution, infectious mortality; safety as prevention of GvHD. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Velardi, Prof, Principal Investigator — Hematology Section, University of Perugia
Locations (1):
- Hematology Section, University of Perugia, Perugia, Perugia, Italy